CLINICAL TRIAL: NCT04452045
Title: Feasibility of a Sleep Intervention for Children With Autism Spectrum Disorder Study
Brief Title: SweetDreams Sleep Study for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UL1TR001872 (NIH)
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder; Insomnia
Keywords: sleep; autism
MeSH Terms: conditions — Autism Spectrum Disorder; Sleep Initiation and Maintenance Disorders; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- SweetDreams (Experimental): Access to a mobile and computer accessible adaptation of existing evidence based sleep interventions.
  Interventions: Device: SweetDreams
- Waitlist Control (No Intervention): Wait list condition with future access to a mobile and computer accessible adaptation of existing evidence based sleep interventions.

INTERVENTIONS:
Device: SweetDreams — SweetDreams is a mHealth adaptation of existing evidence-based sleep interventions. It is a user friendly and developmentally appropriate modularized 4-week web-based intervention available on computer, tablet or mobile phones.
  Arms: SweetDreams

SUMMARY:
This proposal will acquire preliminary data on the feasibility and effectiveness of an innovative and scalable strategy for improving access to effective sleep health care for preschool-aged children with Autism Spectrum Disorder (ASD). The investigators will develop and test an on-line delivery adaptation of the existing behavioral sleep interventions for preschool aged children.

DETAILED DESCRIPTION:
Access to effective treatments for sleep disorders is a persistent challenge. This is due to the lack of trained clinicians as well as caregiver resources to seek out and utilize such critical services. The SweetDreams intervention will solve this problem with on-line delivery of educational materials and treatment strategies for an evidence-based intervention. It will be readily available to caregivers at any time and through multiple outlets such a computer, tablet, and telephone, modes of delivery favored by and effective for parents of children in this age group.

This adaptation will address key challenges to sleep health care for children with ASD: (1) Learning differences of children with ASD by incorporating intervention principles from the TEACHH model; (2) Overcome the challenge of treatment access due to the limited number of qualified providers by developing didactic videos for online and mobile device delivery (referred to as SweetDreams); and, (3) Responding to the NIH emphasis on developing "more effective interventions…by targeting interventions to the identified needs of community members," SweetDreams will use a dynamic process involving extensive collaboration with children, parents, developmental pediatricians, and other experts on youth with ASD.

ELIGIBILITY:
Inclusion Criteria:

* have poor sleep health
* have a diagnosis of ASD

Exclusion Criteria:

* any regular sleep medication use (this does not include occasional over the counter sleep aid)
* known sleep apnea
* unstable major medical conditions (e.g. severe asthma, diabetes).

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Asarnow, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SweetDreams | Waitlist Control
Started | 9 | 11
Completed | 7 | 5
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SweetDreams | Waitlist Control | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: months] | 46.11 (6.74) | 46.27 (10.9) | 46.2 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 6 | 9 | 15
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 2 | 2 | 4
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Children's Sleep Habits Questionnaire (CSHQ)
Description: Validated questionnaire; total score range between 33 and 99, with higher numbers representing more sleep problems
Time Frame: baseline to end of treatment (average exposure 1 month)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SweetDreams | Waitlist Control
Number analyzed (Participants) | 9 | 11
units on a scale | -8.78 (12.3) | -.59 (12.7)

2. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI)
Description: Validated questionnaire; total score range between 0 and 21, with higher numbers representing worse sleep quality
Time Frame: baseline to end of treatment (average exposure 1 month)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SweetDreams | Waitlist Control
Number analyzed (Participants) | 9 | 11
units on a scale | -3.36 (4.17) | .24 (3.99)

ADVERSE EVENTS:
Time Frame: baseline to end of treatment (average exposure 1 month)
Arm/Group | SweetDreams | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT04452045/Prot_SAP_ICF_001.pdf